CLINICAL TRIAL: NCT02651766
Title: Randomised Controlled Trial on the Influence of Cupping Massage on Pain Intensity and Sensory Mechanical and Pain Thresholds in Patients With Chronic Non Specific Neck Pain
Brief Title: The Effects of Cupping Massage in Patients With Chronic Neck Pain - A Randomized Controlled Trial
Acronym: SKM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universität Duisburg-Essen (Other)
Responsible Party: Principal Investigator, Romy Lauche, Principle investigator, Universität Duisburg-Essen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-3987-BO
Record Dates: First submitted 2016-01-07; First posted 2016-01-11 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: Neck Pain; Mechanical/Motor Problems With Neck and Trunk
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Waiting List control group (No Intervention): No treatment within the study period, were allowed to continue physiotherapy and medication. Were offered the treatment after finishing the study
- Cupping massage treatment (Experimental): Received the 5 cupping treatments, application twice a week on the upper back and neck
  Interventions: Procedure: Cupping massage

INTERVENTIONS:
Procedure: Cupping massage — Using suction on the skin by means of glass cups, and moving the cups after applying massage oil on the skin
  Other Names: Moving cupping treatment
  Arms: Cupping massage treatment

SUMMARY:
The study aims to investigate the influence of 5 cupping massage treatments on chronic non specific neck pain. 50 patients with neck pain are randomised into cupping treatment and waiting list control group. Before and after the intervention the investigators evaluate the neck pain (VAS), the neck related disability (NDI), pain on movement (POM) and the quality of life (SF36) and safety. To investigate neurophysiological effects of cupping the investigators also measure mechanical detection threshold (MDT), vibration detection threshold (VDT) and pressure pain threshold (PPT) and the two point discrimination threshold at pain related and control areas.

The treatment group receives 5 cupping treatments over a period of 3 weeks.

DETAILED DESCRIPTION:
see above

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 75
* permanent neck pain for at least three months in a row
* a minimum of 40mm of neck pain on a 100mm visual analogue scale (VAS)

Exclusion Criteria:

* neck pain caused by trauma, inflammatory or malignant disease, by congenital malformation of the spine or if pain was accompanied by radicular symptoms such as radiating pain, paresis, prickling or tingling.
* invasive treatments within the last 4 weeks, surgery to the spine within the last year, corticosteroid or opioid treatment.
* serious acute or chronic organic disease such as diabetes or cancer, mental disorders, pregnancy, and haemorrhagic tendency or anticoagulation treatment.
* non steroidal pain medication and physiotherapy were allowed if the treatment regimen was not altered for four weeks before and continued during the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-05; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 3 weeks
  100mm Visual Analogue Scale from 0mm 'no pain' to 100mm 'maximal pain'

SECONDARY OUTCOMES:
Pain on movement (POM) | 3 weeks
  100mm Visual Analogue Scale from 0mm 'no pain' to 100mm 'maximal pain' Intensity rated for 6 movement directions flexion, tension, and rotation
Neck disability index | 3 weeks
  NDI measures neck pain complaints (Vernon und Mior 1991)
Quality of Life SF-36 | 3 weeks
  the sf-36 is a short form health survey consisting of 8 scales to measure functional health and wellbeing (Bullinger & Kirchberger 1998)
mechanical detection threshold MDT | 3 weeks
  by von Frey filaments to measure perception threshold for light touch (Rolke, Pain, 2006)
vibration detection threshold VDT | 3 weeks
  with a tuning fork to measure perception threshold for vibration (Rolke, Pain, 2006)
pressure pain threshold PPT | 3 weeks
  with a pressure gauge algometer to determine threshold for painful pressure (Rolke, Pain, 2006) on the area of maximal neck pain, the adjacent and hand and foot
Adverse events | 3 weeks
  Number of patients with adverse events
two point discrimination threshold | 3 weeks
  using a pair of circles, determining the distance necessary between those to perceive them as separate sensations

CONTACTS AND LOCATIONS:
Overall Officials: GUstav Dobos, Prof MD, Principal Investigator — University of Duisburg-Essen, Chair of Complementary and Integrative Medicine
Locations (1):
- Knappschaftskrankenhaus, Essen, North Rhine-Westphalia, Germany

REFERENCES:
- [Background] Saha FJ, Schumann S, Cramer H, Hohmann C, Choi KE, Rolke R, Langhorst J, Rampp T, Dobos G, Lauche R. The Effects of Cupping Massage in Patients with Chronic Neck Pain - A Randomised Controlled Trial. Complement Med Res. 2017;24(1):26-32. doi: 10.1159/000454872. Epub 2017 Feb 15. PMID 28219058
- [Result] Schumann S, Lauche R, Hohmann C, Zirbes T, Dobos G, Saha FJ. [Development of lipoma following a single cupping massage - a case report]. Forsch Komplementmed. 2012;19(4):202-5. doi: 10.1159/000341869. Epub 2012 Aug 20. German. PMID 22964987
- [Result] Schumann S, Lauche R, Irmisch G, Hohmann C, Rolke R, Saha F, Cramer H, Choi KE, Langhorst J, Rampp T, Dobos G, Musial F. The effects of 5 sessions of cupping massage on chronic non-specific neck pain: A randomized controlled pilot study. BMC Complementary and Alternative Medicine, 2012, 12 (Supplement 1): 80.